CLINICAL TRIAL: NCT02577770
Title: A Single Center, Double Blind, Randomized, Parallel-group Study to Assess the Effect of 200mg Caffeine,400mg Caffeine and Decaffeinated on Acupuncture Analgesia With the Human Pain Model
Brief Title: The Effect of Caffeine on Acupuncture Analgesia With the Human Pain Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Collaborators: University of Leipzig (Other); Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2014TD0018
Record Dates: First submitted 2015-09-12; First posted 2015-10-16 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Pain
Keywords: Acupuncture; caffeine; pain
MeSH Terms: conditions — Pain | interventions — Acupuncture Therapy; Caffeine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 200mg caffeine plus acupuncture (Experimental): In healthy subjects
  Interventions: Device: acupuncture; Dietary Supplement: 200mg caffeine
- 400mg caffeine plus acupuncture (Experimental): In healthy subjects
  Interventions: Device: acupuncture; Dietary Supplement: 400mg caffeine
- Decaffeinated plus acupuncture (Placebo Comparator): In healthy subjects
  Interventions: Device: acupuncture; Dietary Supplement: Decaffeinated

INTERVENTIONS:
Device: acupuncture — therapeutic acupuncture treatment with actual needles
Dietary Supplement: 200mg caffeine — 8g coffee, po
  Arms: 200mg caffeine plus acupuncture
Dietary Supplement: 400mg caffeine — 16g coffee, po
  Arms: 400mg caffeine plus acupuncture
Dietary Supplement: Decaffeinated — decaffeinated coffee, po
  Arms: Decaffeinated plus acupuncture

SUMMARY:
This is a single center, double blind, randomized, parallel-group study to assess the effect of 200mg caffeine,400mg caffeine and decaffeinated on acupuncture analgesia with the human pain model.

DETAILED DESCRIPTION:
Aim: To evaluate the effect of caffeine on acupuncture analgesia with the human pain model.

Design: Double blind, randomized controlled trial will be performed in Chengdu. The study including two pain models : Potassium pain model and Capsaicin pain model. Both models including the following several groups: 200mg caffeine group, 400mg caffeine group, and decaffeinated group. Participants will be randomly assign to the three groups. Each participants will receive coffee drinking and acupuncture intervention. Each subjects of the Potassium pain model will receive be measured the pain at baseline, 30 minutes after drinking coffee, 10, 20, 30 minutes during acupuncture and 30 minutes after acupuncture intervention completed. Blood samples will be collected at baseline, 30 minutes after drinking coffee, 30 minutes during acupuncture and 30 minutes after acupuncture intervention completed. Each subjects of the capsaicin pain model will be measured the spontaneous pain with VAS scale and the area of hyperalgesia with Von Frey hair at the time of 5 minutes after topical application of capsaicin , 30 minutes after drinking coffee, 10, 20, 30 minutes during acupuncture and 30 minutes after acupuncture intervention completed. Blood samples will be collected at the time of 5 minutes after topical application of capsaicin, 30 minutes after drinking coffee, 30 minutes during acupuncture and 30 minutes after acupuncture intervention completed.

ELIGIBILITY:
Inclusion Criteria:

* Age of a subject is between 18 and 40 years old, male or female
* No known active ongoing disease, in good general health, with a BMI ranging from 18 to 30 kg/m2
* No history of mental disorders,infectious diseases and bleeding disorders. No history of allergic reaction. Females who are not pregnant, lactating, of child-bearing potential, or have no a pregnancy plan within 3 months
* No smoking, drinking alcohol
* No intake of beverage, food and alcohol ,which contains caffeine at least two hours
* No use of any of the methyl purine drugs. No use of any of the drugs ,which can affect the half-life of caffeine, such as: cimetidine, steroids, growth hormone, etc
* No previous experience with acupuncture or other related treatments within 3 days
* Reliable, cooperative, and of adequate intelligence to record the requested information on the questionnaire form
* Informed consent form must be signed by subjects

Exclusion Criteria:

* Subject with serious blood, heart, liver, kidney disease, digestive, or hematopoietic system disease
* Subject with serious mental disorders, infectious diseases and bleeding disorders. Subject has a history of allergic reaction. Females who are pregnant, lactating, of child-bearing potential, or have a pregnancy plan within 3 months;
* Prior use of any type of analgesic drugs before study within 5 half-lives of the drugs
* Use of any of the methyl purine drugs. Use of any of the drugs, which can affect the half-life of caffeine, such as: Sympathomimetic drugs, theophylline drugs , α or β-blockers drugs, and any antihypertensive drugs, etc
* Ingestion of any caffeine-containing beverage, food or alcohol 6 hours or less before study
* Subject has a previous experience with acupuncture or other related treatments within 7 days
* Suffered from medical or psychiatric disorders that prevented them from participating in the study
* Subject who belongs to acupuncture-phobia

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Change of pain threshold will be measured with Potassium Pain Tester for potassium pain | Baseline, 30 minutes after drinking coffee,10,20,30 minutes during acupuncture and 30 minutes after acupuncture intervention completed
Change of pain will be measured with Visual Analog Scale for capsaicin pain | 5 minutes after topical application of capsaicin , 30 minutes after drinking coffee, 10, 20, 30 minutes during acupuncture and 30 minutes after acupuncture intervention completed.
Change of pain will be measured with Von Frey Hair for capsaicin pain | 5 minutes after topical application of capsaicin , 30 minutes after drinking coffee, 10, 20, 30 minutes during acupuncture and 30 minutes after acupuncture intervention completed.

SECONDARY OUTCOMES:
The concentration of caffeine in plasma measured by high performance liquid chromatography in both models | one day after the study( blood samples were collected at Baseline, 30 minutes after drinking coffee,30 minutes during acupuncture and 30 minutes after acupuncture intervention completed.
The concentration of adenosine in plasma measured by high performance liquid | one day after the study( blood samples were collected at Baseline, 30 minutes after drinking coffee,30 minutes during acupuncture and 30 minutes after acupuncture intervention completed.

CONTACTS AND LOCATIONS:
Locations (1):
- Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan, China